CLINICAL TRIAL: NCT04792801
Title: Evaluation of PET TDM FDG-Choline as a Decision-making Tool for Routine Care on Inclusion on the Liver Transplant List for Hepatocellular Carcinoma
Brief Title: PET TDM FDG-Choline as a Decision-making Tool for Routine Care on the Liver Transplant List for HCC
Acronym: TEP CARE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_34; 2020-A000998-31 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma; Liver Transplant
Keywords: Hepatocellular carcinoma; Liver transplantation; PET CT, Fluorodeoxyglucose; Fluorodeoxyglucose; Choline
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HCC and whose liver transplant plan has been validated: Prospective inclusion of patients who are candidates for a transplant for CHC at the University Hospital of Lille and Rouen whose transplant project has been validated with a AFP score ≤ 2.
  The systematic performance of a PET-CT with FDG and a PET-CT with Choline in all patients. At the end of the entire assessment, the patients will be (or not) registered on the transplant list and, for the patients registered on the list, a follow-up will be carried out at the level of a specialized transplant consultation every 3 months at during which the alphafoetoprotein dosage and abdominal imaging will be updated, until liver transplantation.
  Interventions: Radiation: PET TDM FDG-Choline

INTERVENTIONS:
Radiation: PET TDM FDG-Choline — Performing an FDG TDM PET and a Choline TDM PET at two different times

SUMMARY:
HCC is the most common malignant liver tumor for which liver transplantation is one of the pivotal curative treatments. The best possible selection of patients who are candidates for transplantation is essential in the current context of a shortage of transplants. Performing a PET CT scan is not currently recommended in the pre-liver transplant workup for HCC. However, PET CT using in a complementary manner the FDG and Choline tracers appears promising in the management of HCC in view of its wide use in oncology and its major diagnostic and prognostic contribution compared to conventional imaging. In order to address this issue, a prospective cohort study including patients from the University Hospital of Rouen and Lille with hepatocellular carcinoma meeting the criteria for indication of liver transplantation validated in SPC will be set up, the main objective of which will be to assess the decision-making contribution of PET TDM FDG and Choline in addition to conventional imaging in the pre-transplant assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient candidate for liver transplantation for hepatocellular carcinoma from the University Hospital of Lille and Rouen, whose therapeutic transplantation project has been validated and having an AFP score ≤ 2 (diagnosis of HCC defined on non-invasive imaging criteria according to the recommendations of EASL-EORTC 2012 or confirmed histologically).
* No opposition to participating in the study.
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient with an AFP score ≥ 3
* Patient contraindicated to PET FDG or Choline.
* Other tumor: Cholangiocarcinoma.
* Diabetes unbalanced HbA1c> 9%, and fasting hyperglycemia (> 2g / L) which does not allow the completion of the PET examination.
* Patient under guardianship or curatorship.
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant candidates for hepatocellular carcinoma, validated in PCR and having an AFP score ≤ 2.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients reclassified for lymph node fixation (N +) and / or extrahepatic extension (M +) after PET TDM FDG-Choline | through study completion an average of 1 year
  Composite endpoint corresponding to the rate of patients reclassified for lymph node fixation (N +) and / or extrahepatic extension (M +) after PET TDM FDG-Choline with a negative standard assessment (thoracic CT, abdominal imaging by CT or MRI) or patient not included on the list due to locally advanced disease not compatible with the graft (AFP score ≥ 3 or infiltrating HCC) not identified by the standard assessment.

SECONDARY OUTCOMES:
Characteristics of PET FDG-Choline PET binding (defined as below) and the degree of tumor differentiation of HCC on the hepatectomy specimen (well differentiated/ moderate differentiation/ undifferentiated): | At time of liver transplantation (comparison of TEP baseline and HCC obtained on the hepatectomy analysis)
  Presence/absence of a double fixation TEP FDG and TEP Choline B. Presence of a single TEP FDG or Choline binding C. No FDG-Choline binding.
Binding intensity (SUV) of PET TDM FDG-Choline and the degree of tumor differentiation of HCC on the hepatectomy specimen (well differentiated/ moderate differentiation/ undifferentiated) | At time of liver transplantation (comparison of TEP baseline and HCC obtained on the hepatectomy analysis
Binding intensity (SUV) of PET TDM FDG-Choline and risk of waiting list dropout for progression of HCC outside transplant criteria based on aFP score | Analysis on the access to liver transplantation after 24 month.
Binding intensity (SUV) of PET TDM FDG-Choline and risk of HCC recurrence in the 5 years after LT | 5 years after transplantation. Screening for HCC recurrence with CT and abdominal scan every 6 month during 5 years.
Binding intensity (SUV) of PET TDM FDG-Choline and the last aFP value before transplantation or WL dropout. | Last aFP value before LT or WL dropout. Maximal estimated time before transplant: 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lassailly, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France